CLINICAL TRIAL: NCT04711759
Title: Postextubation High-flow Nasal Cannula Versus Standard Oxygen Therapy in Critically Ill Patients: a Physiologic Randomized Crossover Study
Brief Title: Physiologic Effects of High-flow Nasal Cannula Versus Standard Oxygen Therapy Postextubation in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 180814001; 1191709 (Other Grant/Funding Number: Fondecyt)
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2021-01

CONDITIONS: Ventilator Weaning
Keywords: High flow nasal cannula

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Analysis of work of breathing and of data derived from Electric impedance tomography will be performed blind to arm assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A: High flow nasal cannula - Standard oxygen therapy (Experimental): Once participants are extubated they will receive one hour of high flow nasal cannula followed by one hour of standard oxygen therapy.
  Interventions: Device: High flow nasal cannula; Device: Standard oxygen therapy
- Sequence B: Standard oxygen therapy - High flow nasal cannula (Experimental): Once participants are extubated they will receive one hour of standard oxygen therapy followed by one hour of high flow nasal cannula.
  Interventions: Device: High flow nasal cannula; Device: Standard oxygen therapy

INTERVENTIONS:
Device: High flow nasal cannula — High flow nasal cannula will be provided through a commercial device (AIRVO2 + Optiflow nasal cannula, Fisher & Paykel), at 50 LPM and at the same FiO2 applied during the spontaneous breathing trial.
Device: Standard oxygen therapy — Standard oxygen therapy will be provided through a Venturi mask and O2 flow will be adjusted to keep the same FiO2 applied during the spontaneous breathing trial.

SUMMARY:
High-flow nasal cannula (HFNC) is a rather novel system to provide oxygen therapy, which provides flows up to 60 liters/minute (LPM) of heated and humidified gas through nasal prongs. HFNC is increasingly being used in patients with acute respiratory failure. In healthy volunteers and in patients with acute respiratory failure it has been shown to induce several effects beyond those expected for a standard oxygen therapy, such as increased carbon dioxide (CO2) clearance and positive airway pressure.

One of the potential indications for HFNC is to facilitate weaning from mechanical ventilation and extubation. As weaning failure is one of the most complex challenges in mechanically ventilated patients, the use of HFNC after extubation, in order to prevent reintubation, has been evaluated in some clinical trials, with promising results. However, the role of HFNC postextubation is still controversial, and information regarding its effects on the pathophysiologic mechanisms of weaning failure is lacking.

The goal of this proposal is to compare the acute physiologic effects of postextubation HFNC versus standard oxygen therapy, in critically ill patients, on relevant mechanisms related to weaning failure: work of breathing, lung function, systemic hemodynamics.

This will be a randomized crossover study which will include critically ill mechanically ventilated patients, who fulfill criteria indicating they may be ready for weaning from mechanical ventilation, and in whom a spontaneous breathing trial (SBT) is planned to determine if they should be extubated. After checking eligibility and obtaining informed consent, patients will be monitored with an esophageal catheter (esophageal / gastric pressures to determine work of breathing, and electric activity of diaphragm to determine neuromechanical coupling), and a noninvasive ventilation monitor (electric impedance tomography to assess global and regional ventilation). Work of breathing, lung function, and systemic hemodynamics will be assessed during the SBT. Inclusion in the study will be confirmed only if they pass the SBT and are extubated. During the first 2 hours after extubation patients will undergo one hour of HFNC and one hour of standard oxygen therapy, with the crossover sequence being randomized previously at the time of inclusion, and with assessments repeated at the end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation (MV) through an orotracheal tube for at least 48 hours
* PaO2 /FiO2 ratio ≤ 300 mmHg
* Potential for weaning as determined in routine daily screening (precipitating cause leading to MV in resolution, adequate oxygenation (PaO2/FiO2 ≥150 mmHg with FiO2 ≤0.4 and PEEP ≤8 cm H2O), arterial pH >7.25, hemodynamic stability (no vasopressors or Noradrenaline ≤0.1 mcg/kg/min), temperature <38°C, presence of inspiratory effort and appropriate spontaneous cough, and the patient is not receiving sedatives and is awake and able to follow simple commands)
* Decision to perform a spontaneous breathing trial by the attending physician

Exclusion Criteria:

* Patients ventilated for decompensated chronic obstructive pulmonary disease
* Contraindications to HFNC, which include abnormalities or surgery of the face, nose, or airway that preclude an appropriate-fitting nasal cannula.
* Contraindications for esophageal balloon catheter insertion (eg. severe coagulopathy, esophageal varices, and history of esophageal or gastric surgery)
* Contraindication for use of electric impedance tomography (eg. Pacemaker)
* Presence of tracheostomy
* Refusal to participate by the attending physician
* Do not resuscitate order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-12-17 (Actual)

PRIMARY OUTCOMES:
Pressure time-product (PTP) per minute (cmH2O x s/min) | 60 minutes after starting high flow nasal cannula or standard oxygen therapy
  PTPmin will be assessed through an esophageal Neurovent catheter.
Delta end-expiratory lung index (EELI) | 60 minutes after starting high flow nasal cannula or standard oxygen therapy
  Delta EELI will be obtained from electric impedance tomography (EIT) and measured relative to the tidal volume.
Brain natriuretic peptide (BNP) plasma levels | 60 minutes after starting high flow nasal cannula or standard oxygen therapy

SECONDARY OUTCOMES:
Pressure time-product per breath (cmH2O x s) | 60 minutes after starting high flow nasal cannula or standard oxygen therapy
  PTP will be assessed through an esophageal Neurovent catheter.
Peak electric activity of the diaphragm (EAdi) | 60 minutes after starting high flow nasal cannula or standard oxygen therapy
  EAdi will be measured in uV through a Neurovent catheter connected to a Servo-i ventilator
Neuroventilatory efficiency | 60 minutes after starting high flow nasal cannula or standard oxygen therapy
  Vt / EAdi (ml / uV)
Neuromechanical efficiency | 60 minutes after starting high flow nasal cannula or standard oxygen therapy
  Ratio of the (Paw-PEEP) divided by EAdi during inspiratory occlusion (cmH2O / uV)
Global inhomogeneity index | 60 minutes after starting high flow nasal cannula or standard oxygen therapy
  index derived from EIT and calculated from the sum of the impedance changes of each pixel with respect to its median (in absolute values), divided by the sum of the impedance values of each pixel
PaO2 / FiO2 | 60 minutes after starting high flow nasal cannula or standard oxygen therapy
  Parameter of oxygen exchange calculated as the ratio of PaO2 / FiO2

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Bruhn, MD, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clínico UC Christus, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Hernandez G, Vaquero C, Gonzalez P, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Colinas L, Cuena R, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Conventional Oxygen Therapy on Reintubation in Low-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Apr 5;315(13):1354-61. doi: 10.1001/jama.2016.2711. PMID 26975498
- [Background] Fernandez R, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Masclans JR, Lesmes A, Panadero L, Hernandez G. High-flow nasal cannula to prevent postextubation respiratory failure in high-risk non-hypercapnic patients: a randomized multicenter trial. Ann Intensive Care. 2017 Dec;7(1):47. doi: 10.1186/s13613-017-0270-9. Epub 2017 May 2. PMID 28466461
- [Background] Mauri T, Turrini C, Eronia N, Grasselli G, Volta CA, Bellani G, Pesenti A. Physiologic Effects of High-Flow Nasal Cannula in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2017 May 1;195(9):1207-1215. doi: 10.1164/rccm.201605-0916OC. PMID 27997805
- [Derived] Basoalto R, Damiani LF, Jalil Y, Bachmann MC, Oviedo V, Alegria L, Valenzuela ED, Rovegno M, Ruiz-Rudolph P, Cornejo R, Retamal J, Bugedo G, Thille AW, Bruhn A. Physiological effects of high-flow nasal cannula oxygen therapy after extubation: a randomized crossover study. Ann Intensive Care. 2023 Oct 18;13(1):104. doi: 10.1186/s13613-023-01203-z. PMID 37851284